CLINICAL TRIAL: NCT06369285
Title: A Phase 2 Study of Alisertib in Combination With Endocrine Therapy in Patients With HR+, HER2-negative Recurrent or Metastatic Breast Cancer
Brief Title: A Study of Alisertib in Combination With Endocrine Therapy in Patients With HR-positive, HER2-negative Recurrent or Metastatic Breast Cancer
Acronym: ALISCA-Breast1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMA-ALI-1201; 2024-511497-79-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hormone Receptor Positive HER-2 Negative Breast Cancer; Metastatic Breast Cancer; Recurrent Breast Cancer
Keywords: Hormone receptor positive (HR+); Human epidermal growth factor receptor 2 negative (HER2-); Recurrent Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Alisertib 50 mg (Experimental): Alisertib with selected endocrine therapy
  Interventions: Drug: Alisertib; Drug: Endocrine therapy
- Alisertib 40 mg (Experimental): Alisertib with selected endocrine therapy
  Interventions: Drug: Alisertib; Drug: Endocrine therapy
- Alisertib 30 mg (Experimental): Alisertib with selected endocrine therapy
  Interventions: Drug: Alisertib; Drug: Endocrine therapy

INTERVENTIONS:
Drug: Alisertib — Alisertib enteric-coated tablets will be taken by mouth twice daily on days 1-3, 8-10, and 15-17 of each 28-day cycle.
  Other Names: PB-8237; MLN8237
Drug: Endocrine therapy — Investigator selected endocrine therapy will be taken in 28-day dosing cycles according to the approved prescribing information.
  1 mg of anastrozole tablet by mouth once daily or
  2.5 mg of letrozole tablet by mouth once daily or
  25 mg of exemestane tablet by mouth once daily or
  20 mg of tamoxifen tablet by mouth once daily or
  500 mg of fulvestrant intramuscular injection on Study Day 1, 15, 29, and once every 28 days thereafter

SUMMARY:
PUMA-ALI-1201 is a randomized, dose optimization, multicenter, Phase 2 study of alisertib administered in combination with endocrine therapy in participants with pathology-confirmed HR-positive/HER2-negative metastatic breast cancer (MBC) following progression on or after at least two prior lines of endocrine therapy in the recurrent or metastatic setting. This study is intended to evaluate the optimal alisertib dose administered in combination with the selected endocrine therapy. The study is also planned to evaluate the efficacy, safety, and pharmacokinetics of alisertib in combination with endocrine and to identify the biomarker-defined subgroup(s) that may benefit most from combined alisertib and endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at signing of informed consent.
* Pathology-confirmed diagnosis of adenocarcinoma of the breast with evidence of recurrent or metastatic disease not amenable to curative therapy.
* Progression on or after treatment with at least two prior lines of endocrine therapy in the recurrent or metastatic setting. a. If metastatic disease recurrence occurs during or within six months of discontinuing adjuvant endocrine therapy, then that endocrine therapy will count as one line of prior therapy.
* Participants must have received a CDK4/6i in combination with endocrine therapy in the recurrent or metastatic setting.
* HR-positive and HER2-negative tumor status reported per local laboratory testing. HR and HER2 testing must be performed consistent with current American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) or European Society of Medical Oncology (ESMO) guidelines:

Exclusion Criteria:

* Treatment with chemotherapy in the recurrent or metastatic setting.
* Prior treatment with an Aurora Kinase A (AURKA) specific-targeted or pan-Aurora-targeted agent, including alisertib, in any setting.

Note: There are additional inclusion and exclusion criteria. The study center will determine if you meet all of the criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Within Dose Subgroup | From date of randomization to first confirmed Complete or Partial Response, whichever came earlier, assessed up to 48 months
  Objective response rate is defined as the percentage of participants demonstrating a confirmed objective response during the study.
Duration of Response (DOR) Within Dose Subgroup | From start date of response (after date of randomization) to first PD, assessed up to 48 months
  Duration of response is measured from the time at which measurement criteria are first met for Complete Response (CR) or Partial Response (PR) (whichever status is recorded first) until the first date of recurrence or progressive disease (PD) or death is objectively documented.
Disease Control Rate (DCR) Within Dose Subgroup | From date of randomization to first confirmed Complete or Partial Response, whichever came earlier, assessed up to 48 months
  Disease control rate is the proportion of participants who achieve overall tumor response (confirmed CR or PR) or Stable Disease (SD) lasting for at least 24 weeks from randomization.
Progression Free Survival (PFS) Within Dose Subgroup | From date of randomization to date of recurrence, progression or death, assessed up to 48 months
  Progression Free Survival (PFS) is measured in months and based on the local tumor assessment. The time interval from the date of randomization until the first date on which recurrence, progression, or death due to any cause, is documented.
Overall Survival (OS) Within Dose Subgroup | From date of randomization to death, assessed up to 48 months
  Overall survival (OS) is defined as the time from randomization to death due to any cause, censored at the last date known alive on or prior to the data cutoff employed for the analysis, whichever was earlier.
Percentage of Participants With Treatment-Emergent Adverse Events (Adverse Events and Serious Adverse Events) in the Enrolled Population | From date of first dose through last dose plus 28 days, assessed up to 48 months
  Treatment emergent adverse events are those events reported on or after the first dose of investigational product and up to 28 days after last dose.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Within Biomarker-Defined Subgroup | From date of randomization to first confirmed Complete or Partial Response, whichever came earlier, assessed up to 48 months
  Objective response rate is defined as the percentage of participants demonstrating a confirmed objective response during the study.
Duration of Response (DOR) Within Biomarker-Defined Subgroup | From start date of response (after date of randomization) to first PD, assessed up to 48 months
  Duration of response is measured from the time at which measurement criteria are first met for CR or PR (whichever status is recorded first) until the first date of recurrence or progressive disease (PD) or death is objectively documented.
Disease Control Rate (DCR) Within Biomarker-Defined Subgroup | From date of randomization to first confirmed Complete or Partial Response, whichever came earlier, assessed up to 48 months
  Disease control rate is the proportion of participants who achieve overall tumor response (confirmed CR or PR) or SD lasting for at least 24 weeks from randomization.
Progression Free Survival (PFS) Within Biomarker-Defined Subgroup | From date of randomization to date of recurrence, progression or death, assessed up to 48 months
  Progression Free Survival (PFS) is measured in months and based on the local tumor assessment. The time interval from the date of randomization until the first date on which recurrence, progression, or death due to any cause, is documented.
Overall Survival (OS) Within Biomarker-Defined Subgroup | From date of randomization to death, assessed up to 48 months
  Overall survival (OS) is defined as the time from randomization to death due to any cause, censored at the last date known alive on or prior to the data cutoff employed for the analysis, whichever was earlier.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Reg Affairs, PV, Medical Affairs and Law Officer, Study Director — Puma Biotechnology, Inc.
Locations (53):
- United States (35):
  - Alabama Oncology, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - MemorialCare Orange Coast Medical Center, Fountain Valley, California
  - City of Hope at Orange County Lennar Foundation Cancer Center, Irvine, California
  - LA Cancer Network, Los Angeles, California
  - UCLA Department of Medicine - Hematology/Oncology, Los Angeles, California
  - University of California San Francisco (UCSF) Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Illinois Cancer Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Oncology Hematology Associates, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cancer Care Specialists, Reno, Nevada
  - University of Rochester Medical Center, Rochester, New York
  - UNC Hospitals, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Ohio State University, Stefanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - Taylor Cancer Research Center, Maumee, Ohio
  - Alliance Cancer Specialists, Horsham, Pennsylvania
  - University of Pennsylvania, Abramson Cancer Center, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh (UPMC), Pittsburgh, Pennsylvania
  - Tennessee Oncology, Greco-Hainsworth Center for Research, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - Virginia Cancer Institute, Richmond, Virginia
- Portugal (4):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil (IPO Lisboa), Lisbon
  - Fundação Champalimaud, Lisbon
  - Hospital CUF Descobertas, Lisbon
  - Instituto Português Oncologia Do Porto, Porto
- Spain (14):
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clínico de Barcelona, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital San Cecilio, Granada
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario de Jaén, Jaén
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Fundación Instituto Valenciano de Oncología (IVO), Valencia
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Puma Biotechnology is committed to sharing clinical trial data and information to help physicians and patients make informed treatment decisions, and to help qualified researchers advance scientific knowledge.
  In accordance with legal and regulatory requirements, Puma publishes study protocol information and clinical study results on clinical trial registries, including ClinicalTrials.gov and EU Clinical Trials Register. Puma also publishes information about clinical studies in peer-reviewed scientific journals and shares data in scientific meetings.
  Puma commits to safeguarding confidentiality and patient privacy throughout the clinical trial data and information sharing process. Any patient-level data will be anonymized to protect personally identifiable information.
  Qualified researchers and study participants may submit requests for other study documentation and clinical trial data to clinicaltrials@pumabiotechnology.com for consideration.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Clinical study documents and clinical trial data may be requested by qualified researchers and study participants for studies that have been completed for at least 18 months, and for which the indication of the drug has been approved in the US and/or EU, as applicable. Requests will be accepted for up to 24 months after the criteria described in this section are met.
Access Criteria: Requestors must provide organizational contact information; a detailed research plan, including outcomes; timeline for completion of the research; qualifications of the research team; funding source; and potential conflicts of interest.
  Puma will not provide access to patient-level data if there is a reasonable likelihood that individual patients could be identified, or in cases where confidentiality or consent provisions prohibit transfer of data or information to third parties. Additionally, Puma will not disclose information that jeopardizes intellectual property rights or divulges confidential commercial information.
URL: https://pumabiotechnology.com/data_sharing_policy.html